CLINICAL TRIAL: NCT05786365
Title: Comparison of Emergence/Dysphoric Reaction Frequency of Using Ketamine at 2 Different Doses in Interventional Sedation and Analgesia
Brief Title: Comparison of Emergence/Dysphoric Reaction Frequency of Using 2 Different Doses Ketamine
Status: Completed | Type: Observational
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, çağrı türkücü, cagriturkucu, Aksaray University Training and Research Hospital
Other Study IDs: cagriturkucu
Record Dates: First submitted 2023-02-22; First posted 2023-03-27 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Sedation Complication
Keywords: Ketamine; Procedural sedation analgesia; Dysphoric reaction; Sedation
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The group given 0.5 mg/kg ketamine: In this group we will give 0.5 mg/kg ketamine and we observe for disphoric reaction
  Interventions: Drug: Ketalar 50 MG/ML Injectable Solution
- The group given 1 mg/kg ketamine: In this group we will give 1 mg/kg ketamine and we observe for disphoric reaction
  Interventions: Drug: Ketalar 50 MG/ML Injectable Solution

INTERVENTIONS:
Drug: Ketalar 50 MG/ML Injectable Solution — Ketamine will be administered to two different groups as 0.5 mg/kg and 1 mg/kg
  Other Names: ketamine hydrochloride

SUMMARY:
The aim of this study is to compare the effect of using different doses of ketamine on producing dysphoric reaction.

DETAILED DESCRIPTION:
Our study is a randomized single-blind observational study. In our study, the effect of producing a dysphoric reaction will be observed by administering ketamine at doses of 0.5 mg/kg and 1 mg/kg to two randomly randomized different groups who presented to our hospital and needed interventional sedation analgesia. For this reason, our patients with an indication for interventional sedation and analgesia will be taken to the observation room and their vital values will be monitored. Two different vascular accesses with at least 18 gauge will be obtained from the two extremities. The patients will be randomized and 0.5 mg/kg IV ketamine will be given to the 1st group. The second group will be given 1 mg/kg IV ketamine. Then, the patients will be recorded in terms of blood pressure, pulse and saturation at the 5th minute, 15th minute and 30th minute. We will give iv ketamine to two different patient groups as 0.5 mg per kilogram in the 1st group and 1 mg per kilogram in the 2nd group and we will observe the patients.We scored the patients between +4 and -5 points on the RASS scale. Patients who were sedated to an extent that they could not be awakened were scored as -5, patients who were dangerously agitated +4, and patients who were awake were scored 0. We considered patients who scored +2 on the Richmond agitation sedation scale as having developed a dysphoric reaction.

ELIGIBILITY:
Inclusion Criteria:

* Glaskow coma scale should be 15
* Inability to speak, read or understand English or Turkish
* Patients needing procedural sedation and analgesia

Exclusion Criteria:

* Patients with active coronary artery disease
* Patients with liver or kidney transplant
* Patients with conditions that change consciousness such as substance intake, alcohol intake
* Patients with advanced COPD or Heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases with an indication for sedation analgesia, who applied to our emergency department, will be included in our study. Indications for interventional sedation and analgesia: Tube thoracostomy insertion, central venous catheter insertion, fracture/dislocation reduction, skin incision repair, arthrocentesis, lumbar puncture, paracentesis, burn debridement, cardioversion
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
To observe a significant difference between the two doses in terms of producing a dysphoric reaction | January 2023-August 2023
  We will give iv ketamine to two different patient groups as 0.5 miligram/kilogram in the 1st group and 1 miligram/kilogram in the 2nd group and we will observe the patients.We scored the patients between +4 and -5 points on the Richmond Agitation and Sedation Scale between -5 to +4. Patients who were sedated to an extent that they could not be awakened were scored as -5, patients who were dangerously agitated +4, and patients who were awake were scored 0. We considered patients who scored +2 on the Richmond agitation sedation scale as having developed a dysphoric reaction.

SECONDARY OUTCOMES:
Efficacy of 0.5 mg/kg and 1 mg/kg IV ketamine | January 2023-August 2023
  We will give iv ketamine to two different patient groups as 0.5 miligram/kilogram in the 1st group and 1 miligram/kilogram in the 2nd group, and and we will evaluate patients in terms of sedation duration and efficacy.We evaluated the efficacy according to whether additional doses were needed, sedation duration, and the ability to perform the procedural procedure.

OTHER OUTCOMES:
Comparision side effect of iv ketamine between 2 different dose group | January 2023-August 2023
  We will give iv ketamine to two different patient groups as 0.5 miligram/kilogram in the 1st group and 1 miligram/kilogram in the 2nd group, and we will observe the patients in terms of the incidence of side effects.We monitored patients for the following side effects:Hypertension(Defined as a systolic blood pressure (SBP) of 140 mm Hg or more),tachycardia (Heart rate of more than 100 beats per minute),diplopia or nystagmus, nausea and vomiting, respiratory depression (apnea occurring over 10 seconds or oxygen saturation falling below 90%)

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Kokulu, M.D., Principal Investigator — Aksaray UTRH
Locations (1):
- Çağrı Türkücü, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No